CLINICAL TRIAL: NCT00899405
Title: EGFR Pathway Mutations in Lung Cancer Patient Tumors and Blood
Brief Title: Studying Tumor Tissue Samples and Blood Samples to Learn More About DNA Changes in Patients With Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 225287; UCD-155; UCD-200412410; CDR0000583056 (Other: UCD)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Lung Cancer
Keywords: lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Archival tissue specimens and blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with lung cancer: Collection of archival tumor specimen at the beginning of the study and collection of blood samples at the beginning of the study and then at regular intervals

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at tumor tissue samples and blood samples to learn more about DNA changes in patients with lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Examine the mutational status of the EGFR pathway in tumor and blood samples from patients with lung cancer.
* Correlate the EGFR pathway mutations in these samples with clinical outcomes of these patients.

OUTLINE: Archived tumor tissue and blood samples are analyzed via PCR to detect EGFR pathway mutations in DNA.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed lung cancer

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* May have received prior EGFR inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2005-05; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mutational status of the EGFR pathway | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Philip C. Mack, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Cancer Center, Sacramento, California, United States

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/studying-tumor-tissue-samples-and-blood-samples-to-learn-more-about-dna-changes-in-patients-with-lung-cancer-705725/